CLINICAL TRIAL: NCT01969981
Title: An Observational, Prospective, Single-center Study of Placement and Confirmation of Peripheral Inserted Central Catheters Tip Position Using a New Electrocardiographic Method
Brief Title: A Study to Assess Placement and Confirmation of Peripheral Inserted Central Catheters Tip Position Using a New Electrocardiographic Method
Acronym: SHERLOCK 3CG
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: SHERLOCK 3CG; 1626789 (Other: CNIL number)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Anesthesia; Intravenous
Keywords: Peripheral Inserted Central Catheter
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PICC placement
  Interventions: Procedure: PICC placement with Sherlock 3CG

INTERVENTIONS:
Procedure: PICC placement with Sherlock 3CG

SUMMARY:
This is a prospective, single center, observational study. Patients who require a Peripheral Inserted Central Catheters (PICC) will constitute the study population.

The purpose of the study is to determine whether Sherlock 3CG, is adequate means for the total placement of PICC and confirmation of tip of PICC placement and if this method can be conducted safely and efficiently.

Patients will be included during a 6-month period as well as they are ambulatory or hospitalized. The patient's routine care will not be modified and only PICC will be assessed in the present study.

PICC placement will be performed using the Site Rite guidance and tip position will be confirmed using the Sherlock 3CG.

The procedure is the same as the routine habits of the operator (nurse or anesthesiologist); the vascular access team already uses the previous device for CVC placement.

Patients won't be followed up in the study.

DETAILED DESCRIPTION:
Our current Central Venous Catheter placement protocol for PICC includes the resort to UltraSonography (US) and requires fluoroscopy and plain radiographies throughout the PICC insertion and until the confirmation of best placement.

This verification is mandatory to avoid the risks, delays and costs of repositioning the tip, but obtaining a fluoroscopy and plain radiographies in operating rooms can be time consuming and exposes the patient, nurses and physicians to radiations.

The use of endocavitary electrocardiogram for tip position confirmation has been developed since 1985 and is now recognized as an alternative method. It has been recognized as the best technique in other indications, such as hemodialysis. It helps to position PICC tip in proximity to the cavoatrial junction. In Europe, Italian and German teams already use this new method.

A new ultrasound machine offering external sensors and Endocavitary ECG guide is now available (Site Rite and Sherlock 3CG - Tip Confirmation System), which allows the installation and proper placement in the same operation. This Sherlock 3CG TCS has already been approved by the Food and Drug Administration in the US and is indicated for PICC tip placement confirmation in adult patients.

This new ECG guidance method will allow the PICC insertion without any radiation in the operating room.

For the moment, according to the local recommendations, French patients will have to continue to perform one post-procedural X-ray to confirm tip position. This exam will be performed in a dedicated room of the radiology unit. But guidance and confirmation of CVC placement only by ECG may provide a faster means of confirmation and eliminates radiation exposure to the patients, nurses and anesthesiologists.

In addition, it would eliminate the costs associated with confirmatory chest X-ray (exam costs and time consumption).

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old patient or older,
* Patient requiring PICC placement in the vascular access unit,
* Patient able to read and understand the French language,
* Patient affiliated with a social security system.

Exclusion Criteria:

* Any contraindication to PICC insertion,
* Patient unable to lie in the supine position
* Patient with a Body Mass Index > 40
* Any medical condition that could change the normal presentation of the P-wave such as arrhythmia, atrial flutter, pace maker with permanent stimulation…

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included as well as they are ambulatory or hospitalized in Centre Leon Berard.
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of PICC placement using the Sherlock 3CG | During the procedure (Day 0)
  Success rate of PICC placement (no need to use radiation or fluoroscopy before the end of the procedure)

SECONDARY OUTCOMES:
Assess the number of punctures in brachial site | During the procedure (Day 0)
  Efficacy of needle guide
Assess the unique punction rate | During the procedure (Day 0)
Assess the number of repositions after procedure closed | During the procedure (Day 0)
Assess pain | During the procedure (Day 0)
  By means of a Verbal Numeric Scale
Assess acute complications rate | During the procedure (Day 0)
  Hemothorax, arterial puncture, etc.
Assess the percentage of patients requiring fluoroscopy | During the procedure (Day 0)
Assess the final radiation rate | During the procedure (Day 0)
  When applicable
Assess the percentage of patients with good placement on the X-Ray | During the procedure (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé ROSAY, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France